CLINICAL TRIAL: NCT07077603
Title: Acceptability and Feasibility of an Online Yoga Programme for Adults With a Functional Neurological Disorder.
Brief Title: The Feasibility and Acceptability of an Online Yoga Program for People With Functional Neurological Disorders
Acronym: YOGA-FUND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24NS004
Record Dates: First submitted 2025-04-15; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Functional Neurological Disorder; Dissociative Seizures; Psychogenic Seizure; Non-Epileptic Seizure
Keywords: dissociative seizure; functional neurological disorder; psychogenic seizure; yoga
MeSH Terms: conditions — Conversion Disorder; Psychogenic Nonepileptic Seizures; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients living with a functional neurological disorder (Experimental): Patients living with a functional neurological disorder receiving a 12 week, twice weekly, small group, online yoga sessions
  Interventions: Other: A12 week, twice weekly, small group, online yoga program

INTERVENTIONS:
Other: A12 week, twice weekly, small group, online yoga program — A 12 week, twice weekly, small group, online yoga program

SUMMARY:
This is a feasibility study to see if it is acceptable and helpful for people living with a functional neurological disorder to receive online group yoga sessions to improve their wellbeing

DETAILED DESCRIPTION:
1. BACKGROUND Functional neurological disorders (FND), previously named as either conversion disorder or somatic symptom disorder, are clinical conditions characterized by involuntary motor and sensory symptoms, for example seizures, paralysis, or a tremor, in the absence of any abnormal pathophysiology. Patients' memory, concentration, and cognition can also be impaired .The two most frequent presenting symptoms are seizure-like episodes, also known as dissociative or psychogenic non-epileptic seizures, or persistent motor effects that resemble a stroke. The current UK prevalence of FND is poorly understood with estimates ranging between 50,000 to 100,000, and an annual new incidence of 8,000. This is likely to be grossly underestimated, as FND is frequently misdiagnosed and thought to be the cause of up to 30% (n=1,444/4,299) of all presentations to neurology clinics and 10-20% of Neurology inpatients at Nottingham University Hospitals. FND is more common in women than men (3:1) and less common in infants than adults . In Nottinghamshire, approximately 100 people with FND seek advice from the neurology services at Nottingham University Hospitals NHS Trust each month either through clinics, telephone, or email. There is a significantly high burden of disability in this patient population, with physical symptoms equivalent to multiple sclerosis or epilepsy, along with anxiety, depression, chronic fatigue and "brain fog". The causes of FND remain unknown. It is difficult to diagnose FND because it cannot be explained as a medical or neurological disease, there is no formal gold standard diagnostic criteria, and there are currently no medical or physiotherapy curative treatments. Overall, the optimal healthcare management of people with FND remains a major challenge.

   The absence of a definitive medical or physiotherapy cure for FND has led to the exploration by the Nottingham University Hospitals clinical team of non-medical approaches to symptom management. Yoga, a holistic physical, mental, and spiritual practice that originates from India, uses repetitive physical postures and stretches (asanas), breathing exercises (pranayama), and meditation (dyana) to improve physical and psychological wellbeing. Yoga has been demonstrated to improve the health related quality of life (HRQOL) in populations aged 60 years and over, and amongst adults with multiple sclerosis and reduce anxiety and depression. Overall, holistic approaches to care view the person as a whole being and consider their social, psychological, and spiritual needs in addition to their physical health needs.

   In December 2023, a systematic search for publications detailing Yoga interventions for people with FND was conducted by the study Chief Investigator. This comprehensive search yielded two conference abstracts detailing the outcomes of case studies (n=3 patients) by the same author reporting improvements in pain, muscle spasms, balance, and anxiety. Thus, there are two research gaps present, namely knowledge (where research findings do not exist) and population (a lack of data pertaining to the population and phenomenon of interest).
2. RATIONALE The World Health Organization define health as being "a state of complete physical, mental and social well-being and not merely the absence of disease and infirmity". People living with FND experience symptoms in all three physical, mental and social well-being domains, accompanied by misunderstanding and stigmatizing behaviour by both members of the public and by healthcare professionals. Although the prevalence of FND is greater than that of multiple sclerosis and has similar symptom severity, both clinical treatment and clinical research opportunities are limited. Recommendations for the construction of an optimum clinical pathway for FND that recognises symptom heterogeneity and the need to integrate physical and psychological health services have been developed by the National Neurosciences Advisory Group. This clinical pathway includes the provision of practical self-management actions for patients. Yoga is a practical activity that can be taught and practiced individually in isolation or in facilitated groups.

In this study, the specific sub-population of people with FND of interest is those who experience psychogenic non-epileptic seizures (PNES), also known as dissociative seizures (DS). Seizures can be differentiated between being epileptic or non-epileptic by recording a seizure on video electroencephalography, or by an expert neurological clinical assessment of the history preceding a seizure, the characteristics of the seizure, and normal electroencephalography patterns during seizures and at baseline.

The association between PNES, and symptoms of depression and anxiety is established. The word yoga means unite, referring to the joining of the mind and body, so is an appropriate interventional approach to consider for this population. An integrative cognitive model of PNES posits that the seizures are linked to sympathetic nervous system activation by chronic stress or factors that compromise inhibitory control processing (a cognitive process that enables individuals to suppress impulses or strong behavioural responses to a stimuli). The Polyvagal Theory explains that feeling psychologically unsafe, even in situations that are objectively safe, unconsciously activates the sympathetic nervous system function, so it follows that this could be a further contributory factor.

An established action-orientated approach to psychotherapy called Acceptance and Commitment Therapy (ACT) comprises six features, one of which is "being mindful in the present moment" . In keeping with the Integrated Care Model (ICM) and Polyvagal Theory, the ACT approach recognises that suppressing emotionally or psychologically painful and difficult experiences is counterproductive and can increase distress. The planned yoga intervention in this study will engage the parasympathetic nervous system, and facilitate calm and reduce stress, thus supporting both the ICM, ACT, and the Polyvagal Theory via three mechanisms. First, the deep relaxation and mindfulness in the Yoga Nidra and Meditation sections are aligned with the ACT and Polyvagal Theories . Secondly, the Bramhari Pranayama (honeybee breathing, or humming) in the Meditation section will directly engage the autonomic nervous system and increase parasympathetic and decrease sympathetic activity. Finally, the group online yoga programme facilitated by an expert yoga practitioner and neurological care registered nurse has been designed to promote a psychologically safe group social space, which will also activate the Polyvagal Theory.

Furthermore, some patients with FND and seizures may also experience long term chronic pain in the form of fibromyalgia, complex regional pain syndrome, or irritable bowel syndrome.

The National Institute of Health and Care Excellence recognise the detrimental long-term effects that prescribed analgesic agents can cause, including addiction, paired with variable evidence of efficacy. In particular, for chronic primary pain, their guidelines emphasize how a person's experience of pain is typically influenced by social and emotional factors, mental health, expectations, beliefs, and biological factors. Thus NICE now recommend non-pharmacological interventions for chronic pain management that include relaxation therapies, group exercise programmes, and social interventions all of which will be met by the planned yoga programme in this feasibility study. Participants' experiences of pain, and any seizure frequency and duration, will be collected during this study. However the primary outcomes measured focus on wellbeing rather than on any physical health metrics.

A 10 week pilot project was introduced at Nottingham University Hospitals NHS Trust in 2022 comprising a once weekly one-to-one online yoga to six patients with FND. The six patients participated in a post intervention focus group and verbally reported universally positive feedback, a reduction in anxiety, improvements in mental well-being, continued use of breathing techniques, and that yoga delivered in group sessions for a longer duration would be of benefit.

Against this background, the proposed single site feasibility study will measure the impact of small group, online yoga on the self-reported health and mental well-being of people with a functional neurological disorder whose primary symptoms are seizure-like episodes.

Although the investigators will capture patients' experiences of pain and any episodes of seizures during the 12 week programme duration, the study will focus on acceptability (acceptable to those delivering and receiving the intervention), and adaptation (adapting a yoga programme content and delivery to the FND patient population).

ELIGIBILITY:
Inclusion Criteria:

* Participants able to give informed consent.
* Aged 18 years and over.
* Participants with a confirmed clinical diagnosis of functional neurological disorder with dissociative seizures.
* Access to WiFi and an electronic device on which to view and participate in the yoga programme.

Exclusion Criteria:

* Participants with severe fatigue that would prevent engagement for the duration of the intervention (assessed by clinical neurology team member).
* Participants who regularly practice yoga i.e., participants who practice each week.
* People with a confirmed concurrent diagnosis of epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The number of participants who fully complete their twice weekly, 12 week online yoga intervention. | This data will be recorded at the end of each participants 12 week planned intervention duration.
  The number of participants who fully complete their twice weekly, 12 week online yoga intervention will be recorded as an indicator of whether the intervention was acceptable to receive and feasible to deliver and receive.

SECONDARY OUTCOMES:
Improvements in participants' self-reported health and well-being measured by the Brief Illness Perceptions Questionnaire. | At baseline before the intervention begins, and between 1 and 14 days following the completion of the intervention.
  This is an eight-item questionnaire in which participants rate each of the health and wellbeing metrics on a scale between 0-10, where higher scores indicate better health and wellbeing outcomes for questions 3,4,7, and higher scores indicate poorer health and wellbeing outcomes for questions 1,2,5,6,8. Participants can also report what they believe has caused their illness.
Improvements in participants' self-reported self-management measured by the Self-Management Assessment Scale. | At baseline before the intervention begins, and between 1 and 14 days following the completion of the intervention.
  This is a ten-item questionnaire in which participants rate each of the self-management metrics on a scale between 0-6, where higher scores indicate better self-management outcomes for all ten questions.
Improvements in participants' self-reported mental wellbeing measured by the Warwick-Edinburgh Mental Wellbeing Scale. | At baseline before the intervention begins, and between 1 and 14 days following the completion of the intervention.
  This is a 14-item questionnaire in which participants rate each of the mental wellbeing metrics on a five-point Likert scale ranging from "none of the time" to "all of the time", where the "all of the time" responses indicate better mental wellbeing outcomes for all fourteen questions.
Improvements in participants' self-reported mental health measured by The Patient Health Questionnaire-9 (PHQ-9). | At baseline before the intervention begins, and between 1 and 14 days following the completion of the intervention.
  This is a ten-item questionnaire in which participants rate each of the nine mental health metrics on a four-point Likert scale ranging from "not at all" to "nearly every day", where the "nearly every day" responses indicate worse mental health outcomes for all nine questions. The last question asks participants to indicate, on a four-point Likert scale ranging from "not difficult at all" to "extremely difficult", if any of the issues in the previous nine questions that they have experienced have led to difficulties at home, at work, or when interacting with other people.
Improvements in participants' self-reported levels of physical pain measured by the British Pain Society Pain Rating Scale. | At baseline before the intervention begins, and between 1 and 14 days following the completion of the intervention.
  This is an six-item questionnaire in which participants rate their experiences of pain on a scale between 0-10, where higher scores for questions 1-5 indicate extreme or distressing pain, and a higher score for question 6 indicates improved pain control.
Improvements in participants' self-reported levels of fatigue measured by the The Functional Assessment of Chronic Illness Therapy (FACIT) scale. | At baseline before the intervention begins, and between 1 and 14 days following the completion of the intervention.
  This is a 13-item questionnaire in which participants rate each of the fatigue metrics on a five-point Likert scale ranging from "not at all" to "very much", where the "very much" responses indicate worse fatigue to questions 1-6 and 9-13, and improvements in fatigue for questions 7 and 8.

IPD SHARING:
Plan to Share IPD: No